CLINICAL TRIAL: NCT00604149
Title: Etude Multicentrique en Population de la susceptibilité génétique à Faire Une Mort Subite
Brief Title: Cardiac AResT And GENEtic
Acronym: CARTAGENE
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C07-35; 2007-A01048-45 (Registry Identifier: IDRCB)
Record Dates: First submitted 2008-01-16; First posted 2008-01-30 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Out-of-hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood to obtain DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: case of out-of-hospital cardiac arrest
- 2: cases of MI
- 3: controls without coronary disease

SUMMARY:
Sudden death is a major problem in industrially developed countries. Despite a decline in ischemic heart disease mortality and the progress has been made in resuscitation, treatment of sudden death victims is frequently unsuccessful. the ideal solution would be to prevent the disease process that causes the initial episode of cardiac arrest. Parental sudden death is an independent risk factor for sudden death. So, detect a gene predisposing to sudden death may help provide better identification of subjects at high risk of cardiac arrest. This research is a genetic study of sudden cardiac death, recruited 2000 subjects in out-of-hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* OHCA
* Aged from 18 to 75 years

Exclusion Criteria:

* Pregnant
* People not free
* Inhospital subjects
* Death by other disease
* Violent death

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all subjects in out-of-hospital cardiac arrest and treated by medical mobil emergency medical care
Sampling Method: Non-Probability Sample
Enrollment: 2332 (Actual)
Dates: Start 2008-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Jouven, PhD, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France